CLINICAL TRIAL: NCT06138899
Title: Enhancing Blood Donation Rates at Schools and Beyond Using Club 25 Blood Donor Program in Malawi: An Implementation Science Study
Brief Title: Enhancing Blood Donation at Schools and Beyond in Malawi
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Malawi Blood Transfusion Services (MBTS) (Unknown); University of North Carolina, Chapel Hill (Other); Ministry of Health, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B10; 5UH3HL152189-04 (NIH)
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Blood Donation

STUDY DESIGN:
Intervention Model Description: Hybrid Type I implementation-science cluster-randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Club 25 (Experimental): Club 25 donation programs will be set up in schools randomized to this arm. Three blood donation events per school year will take place at study schools. Each donation event will be preceded by a motivational talk intended to inform students of the importance of blood donation and encourage students to donate blood. Donation events and motivational talks will be planned and conducted by the Malawi Blood Transfusion Services (MBTS).
  Interventions: Other: Club 25
- Standard procedures (No Intervention): Schools in this arm will not take part in a Club 25 donation program. Three blood donation events per school year will take place at study schools. Each donation event will be preceded by a motivational talk intended to inform students of the importance of blood donation and encourage students to donate blood. Donation events and motivational talks will be planned and conducted by the Malawi Blood Transfusion Services (MBTS).

INTERVENTIONS:
Other: Club 25 — The Club 25 donation program will involve students pledging to donate blood 25 times in their lifetime. In order to achieve this objective, students also pledge to lead a healthy lifestyle, to avoid acquiring HIV and other TTIs and to continue donating blood after leaving school. The Club 25 donation program includes activities in-between blood donation events as well as peer leadership and peer education in schools and in communities.
  Arms: Club 25

SUMMARY:
First developed in Zimbabwe, Club 25 is an initiative to promote blood donation among young people, who present a low-risk population for the spread of transfusion transmissible infections (TTIs). Club 25 members in Malawi make a pledge to donate blood 25 times during their lifetime. The primary aim of this study is to compare a Club 25 donation program to the current standard procedures for student blood donor recruitment in 30 secondary schools in Malawi. Roughly half of the schools will be randomly assigned to a Club 25 intervention and the study will collect data on student blood donations in all 30 schools for three school years. Upon completion of data collection the rate of student blood donation will be compared between the intervention schools and the non-intervention schools.

DETAILED DESCRIPTION:
Recognizing the role of youth in blood donation, Zimbabwe, a country with similar demographics to Malawi, developed "Club 25" in 1989 as a means to encourage regular blood donation among the youth. Club 25 donation programs involved students pledging to donate blood 25 times in their lifetime. In order to achieve this objective, students pledged to lead a healthy lifestyle, to avoid acquiring HIV and other TTIs and to continue donating blood after leaving school. Club 25 in Zimbabwe demonstrated a consistent drop in HIV infection among donors over time and managed to minimize blood shortages during school holidays.

This is a hybrid Type I implementation science cluster randomized clinical trial comparing an enhanced Malawian-tailored school-based Club 25 donation program to the current standard procedures (SP) for student blood donor recruitment in 30 secondary schools in Malawi. This study will be conducted for 3 years, with additional 6 months start-up and 6-month data analysis/write up (total activity period will be 4 years). The total sample size is 11,492 per year. A minimum of 5746 student voluntary non-numerated blood donors (VNRBD) from each arm (15 schools with standard procedures for blood donor recruitment (SP) and 15 Club 25 schools) will be recruited annually. Focus group discussions, in-depth interviews, and key informant interviews will be conducted with a minimum of 400 participants including student VNRBDs, key informants, and community stakeholders. Schools will be stratified by Malawi Blood Transfusion Service regional office sites (South, East, Centre, North).

ELIGIBILITY:
Inclusion Criteria:

* At least 16 years old and enrolled in a secondary school

Exclusion Criteria:

* Under 16 years of age or not enrolled in a secondary school

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35000 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Donation rate | 36 months
  Blood donation rate per year among secondary students

SECONDARY OUTCOMES:
Students who donated at least once | 36 months
  Proportion of the students who donated blood at least once during the course of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Malawi Blood Transfusion Services, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No
The BLOODSAFE project is committed to quickly sharing results and data. Papers will be submitted summarizing the primary results of the BLOODSAFE studies once the analysis is complete. These results will be published in major scientific journals and presented at scientific meetings.